CLINICAL TRIAL: NCT04697511
Title: A Phase I, Single-Sequence, Open-Label, Single- and Multiple-Dose Study of the Effect of Evobrutinib on Midazolam Pharmacokinetics in Healthy Participants
Brief Title: Drug-drug Interaction Study of Evobrutinib With Midazolam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MS200527_0063; 2020-003668-13 (EudraCT Number)
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: Midazolam; Cytochrome P450; Autoimmune disorders; Inflammatory disorders; Sedative-hypnotic
MeSH Terms: conditions — Autoimmune Diseases | interventions — Midazolam; evobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midazolam and/or M2951 (Experimental)
  Interventions: Drug: Midazolam; Drug: M2951

INTERVENTIONS:
Drug: Midazolam — Participants will receive single oral dose of midazolam on Days 1, 3 and 13 under fed conditions.
Drug: M2951 — Participants will receive multiple oral doses (twice daily) of M2951 on Day 3 to Day 13 under fed conditions.
  Other Names: MSC2364447C; Evobrutinib

SUMMARY:
The study will investigate the effect of single dose and multiple doses of M2951 on midazolam Pharmacokinetics (PK) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as determined by medical evaluation, including no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion
* Participants have a body weight within 50.0 and 100.0 kilograms [kg] (inclusive) and body mass index within the range of 19.0 and 30.0 kilograms per square meter [kg/m^2] (inclusive)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders, as determined by medical evaluation
* Individuals with diagnosis of hemochromatosis, Wilson´s disease, alpha 1 antitrypsin deficiency, or any other chronic liver disease including Gilbert's disease will be excluded from the study
* Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to Screening
* History of any malignancy
* History of chronic or recurrent acute infection or any bacterial, viral, parasitic or fungal infections within 30 days prior to Screening and at any time between Screening and admission, or hospitalization due to infection within 6 months prior to Screening
* History of shingles within 12 months prior to Screening
* History of drug hypersensitivity, ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients; history of serious allergic reactions leading to hospitalization or any other hypersensitivity reaction in general, which may affect the safety of the participant and/or outcome of the study per the Investigator's discretion
* History of alcoholism or drug abuse within 2 years prior to Screening, or positive for drugs of abuse, nicotine/cotinine or alcohol by the laboratory assays conducted during Screening and Day -1
* History of residential exposure to tuberculosis, or a positive QuantiFERON® test within 4 weeks prior to or at the time of Screening
* Administration of live vaccines or live-attenuated virus vaccines within 3 months prior to Screening
* Moderate or strong inhibitors or inducers of Cytochrome P450, family 3, subfamily A (CYP3A4/5) within 4 weeks prior to the first administration of study intervention
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUC0-inf) of Midazolam | Pre-dose through 24 hours postdose on Days 1, 3 and 13
Maximum Observed Plasma Concentration (Cmax) of Midazolam | Pre-dose through 24 hours postdose on Days 1, 3 and 13

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Day 14
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) by Severity | Up to Day 14
Number of Participants with Clinically Significant Change From Baseline in Laboratory Parameters, Vital Signs and 12-Lead Electrocardiogram (ECG) Findings | Up to Day 14
  Number of participants with clinically significant change from baseline in laboratory parameters, vital signs and 12- lead ECG findings will be reported.
Area Under the Plasma Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUC0-inf) of 1-hydroxymidazolam | Pre-dose through 24 hours postdose on Days 1, 3 and 13
Maximum Observed Plasma Concentration (Cmax) of 1-hydroxymidazolam | Pre-dose through 24 hours postdose on Days 1, 3 and 13
Time to Reach Maximum Plasma Concentration (tmax) of Midazolam and 1-hydroxymidazolam | Pre-dose through 24 hours postdose on Days 1, 3 and 13
Apparent Terminal Half-life (t1/2) of Midazolam and 1-hydroxymidazolam | Pre-dose through 24 hours postdose on Days 1, 3 and 13
Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t) of Midazolam and 1-hydroxymidazolam | Pre-dose through 24 hours postdose on Days 1, 3 and 13
Apparent Total Body Clearance (CL/F) of Midazolam | Pre-dose through 24 hours postdose on Days 1, 3 and 13
Apparent Volume of Distribution (Vz/F) of Midazolam | Pre-dose through 24 hours postdose on Days 1, 3 and 13

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0063
- See also: Medical Information Location Map - Med Info Contacts — http://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html